CLINICAL TRIAL: NCT00511134
Title: A Placebo-Controlled, Randomized Trial of Eszopiclone for the Treatment of Bupropion- and Abstinence-Related Insomnia During Smoking Cessation
Brief Title: Study of Lunesta Versus Placebo for Sleep Problems Related to Smoking Cessation and Zyban
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study has been terminated due low recruitment of participant population.
Sponsor: Yale University (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0609001866; ESRC099
Record Dates: First submitted 2007-08-01; First posted 2007-08-03 (Estimated); Results first posted 2009-12-04 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Insomnia; Nicotine Dependence
Keywords: insomnia; nicotine dependence; smoking; smoking cessation; zyban
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Tobacco Use Disorder; Smoking; Smoking Cessation | interventions — Eszopiclone; Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zyban + Lunesta (Experimental): Zyban (150 mg qd x 7 days then 150 mg bid x 6 weeks) + Lunesta (3 mg qd x 6 weeks)
  Interventions: Drug: Eszopiclone; Drug: Bupropion
- Zyban + Placebo (Placebo Comparator): Zyban (150 mg qd x 7 days then 150 mg bid x 6 weeks) + placebo (1 pill per day x 6 weeks)
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Eszopiclone — eszopiclone (lunesta) - 3 mg qd x 6 weeks, oral capsule
  Other Names: Lunesta
  Arms: Zyban + Lunesta
Drug: Bupropion — bupropion SR in oral capsule will be begun at the beginning of week 1 (150 mg qd x 7 days) with an increase to the full dose (150 mg bid x 6 weeks) at the beginning of week 2.
  Other Names: Zyban

SUMMARY:
Objectives:

The primary objective of this study is to determine the efficacy of eszopiclone at treating sleep problems related to withdrawal from nicotine in healthy smokers attempting smoking cessation.

Sleep disturbances are a significant problem for smokers who are trying to quit smoking. Smokers may be more likely to have sleep problems and both nicotine withdrawal and agents used to aid smoking cessation (e.g., pharmacotherapies) may disrupt sleep. Lunesta (eszopiclone) is a medication that has been approved by the FDA to treat insomnia. Eszopiclone's efficacy for treating insomnia makes it a promising agent for treating nicotine withdrawal-related symptoms of sleep disturbance.

This study will be 7 weeks duration. All participants will begin taking Zyban at the beginning of week 1 and will be asked to try to quit smoking at the beginning of week 2. Participants will also begin to take Lunesta or matched placebo (3 mg qd x 6 weeks) on the target quit date at the beginning of week 2. All subjects will receive eight (8) weekly sessions of brief individual supportive smoking cessation counseling.

Hypothesis:

It is hypothesized that significantly fewer sleep problems will be reported by participants taking Lunesta as compared to placebo. Specifically, it is expected that participants taking Lunesta will report less difficulty falling and staying asleep, higher sleep quality, and less insomnia-related fatigue and distress than participants taking placebo.

ELIGIBILITY:
Inclusion Criteria:

* Are between ages 18-65 years old.
* Meet DSM-IV criteria for nicotine dependence.
* Smoke at least 15 cigarettes (3/4 pack) daily (averaged over 1 week, in the past 1 month) and have an expired breath CO level > 10.
* At the time of initial evaluation, are motivated to quit smoking in the next 30 days.
* Receive a score of ≥ 10 on the Insomnia Severity Index (ISI)
* Have the capacity to give informed consent, and are English-speaking.

Exclusion Criteria:

* Are taking an over-the-counter or prescription medications that are known to affect sleep.
* Are taking medications contraindicated for use with eszopiclone or bupropion including: Ketoconazole, Itraconazole, Clarithromycin, Erythromycin, Nefazodone, Troleandomycin, Ritonavir, Nelfinavir, Trazodone, and Methadone.
* Are using any over-the-counter analgesics that contain caffeine.
* Have serious medical disorders that may make participation in the trial unsafe.
* Are physiologically dependent on and/or abusing alcohol or other drugs of abuse (e.g., cocaine, opiates, benzodiazepines, etc.) in the past 6 months prior to randomization into the trial.
* Consume greater than 1 alcoholic beverage per day or greater than 7 alcoholic drinks per week.
* Meet DSM-IV criteria for a current diagnosis of major depressive disorder, panic disorder or post-traumatic stress disorder, or a current or past history bipolar disorder, schizophrenia, or anorexia or bulimia nervosa. Have a past history of major depression, with historical evidence of suicidal or homicidal behavior, or psychotic symptoms.
* Have the presence of suicidal or homicidal ideation, or significant impairment of social or occupational functioning, either at study baseline during the evaluation process, or during participation in the trial.
* Are from the same household as another study participant.
* A history of seizures of any etiology.
* A history of hypersensitivity to bupropion or Lunesta (eszopiclone).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea H. Weinberger, Ph.D., Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Greater New Haven area and surrounding communities through targeted television, radio, and newspaper ads, fliers, and referrals from clinicians. Recruitment occurred between July of 2007 and October of 2008. Approximately 900 phone screens and 12 in-person screens were completed during the course of the study.
Pre-assignment Details: Major reasons for exclusion at phone screen were report of no sleep problems, use of illegal substances, psychiatric or medical exclusions, and low smoking. Major reasons for exclusion during the in-person screening process included withdrawal of informed consent, alcohol or illicit drug use, and low smoking.
Groups:
- Zyban + Lunesta: Bupropion SR (Zyban; 150 mg qd x 7 days, then 150 mg bid x 6 weeks) and Eszopiclone (Lunesta; 3 mg qd x 6 weeks)
- Zyban + Placebo: Bupropion SR (Zyban; 150 mg qd x 7 days, then 150 mg bid x 6 weeks) and placebo pill (1 pill per day x 6 weeks)
Period: Overall Study
Arm/Group | Zyban + Lunesta | Zyban + Placebo
Started | 1 | 3
Completed | 1 | 1
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zyban + Lunesta | Zyban + Placebo | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Level of Insomnia as Measured by the Insomnia Severity Index
Description: Insomnia Severity Index (ISI): 13-item self-report measure which examines symptoms of insomnia, consequences of insomnia, and subjective distress related to sleep problems. Subjects rate the symptoms and consequences of insomnia on a 5 point Likert scales. For example, subjects are asked to rate the severity of their insomnia (e.g., difficulty falling asleep from 0=none to 4=very severe). Scores on the first 7 items are summed for a total insomnia score ranging from 0-28.
Time Frame: 6 weeks after target smoking quit date
Population: Baseline descriptive data was examined for the 4 participants. Outcome measures were available for 2 participants. Due to the small number of participants, statistical comparisons were not able to be performed.
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | Zyban + Lunesta | Zyban + Placebo
Number analyzed (Participants) | 1 | 1
Units on a Scale | 11 (0) [11 to 11] | 5 (0) [5 to 5]
Statistical Analysis 1: Comparison: Zyban + Lunesta vs Zyban + Placebo; It was hypothesized that the Zyban+Lunesta group would report lower ISI scores at end of trial than the Zyban+Placebo group; Test type: Superiority or Other; p < 0.05, Descriptive data

2. Secondary Outcome: Smoking Abstinence as Measured by Self Reported Smoking and Confirmed by CO Level
Description: Endpoint abstinence will be defined as 0 cigarettes over the seven days prior to the subject's Timeline Follow-Back evaluation at the end of week 7 (end of trial) and a Carbon Monoxide (CO) level ≤ 5.
Time Frame: 6 weeks after target smoking quite date
Measure: Number; unit: participants
Arm/Group | Zyban + Lunesta | Zyban + Placebo
Number analyzed (Participants) | 1 | 3
participants | 1 | 1
Statistical Analysis 1: Comparison: Zyban + Lunesta vs Zyban + Placebo; It is predicted that subjects taking eszopiclone will be more likely to report abstinence at trial endpoint than those taking placebo; Test type: Superiority or Other; p < 0.05, Fisher Exact; Degrees of freedom=1

ADVERSE EVENTS:
Time Frame: 1 year, 3 months
Description: weekly questionnaire
Arm/Group | Zyban + Lunesta | Zyban + Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less